CLINICAL TRIAL: NCT07320716
Title: A Phase 2, Open-Label, Single-Center, Long-Term Immunogenicity Follow-Up Study of the GVGH altSonflex1-2-3 Shigella Vaccine 1, 2 and 3 Years After Vaccination in African Children
Brief Title: Long-Term Immunogenicity of the altSonflex1-2-3 Shigella Vaccine in African Children
Acronym: H06_04TP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 223136
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Diarrhoea
Keywords: Shigella sonnei; Shigella flexneri; Shigella vaccine; altSonflex1-2-3; Shigelllosis
MeSH Terms: conditions — Diarrhea | interventions — Meningococcal Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Tetanus Toxoid; Hepatitis B Vaccines

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- H06_01TP Study_Infants_Selected dose (Experimental): Infants who received 3 doses of the altSonflex1-2-3 vaccine on Day 1, Day 85, and Day 253 in the H06_01TP parent study.
  Interventions: Biological: AltSonflex1-2-3
- H06_01TP Study_ ST2_Infants_Control (Active Comparator): Infants who received 2 doses of the Menveo vaccine on Day 1 and Day 85, and 1 dose of the Infanrix hexa vaccine on Day 281 in the H06_01TP parent study.
  Interventions: Biological: Menveo; Biological: Infanrix hexa
- H06_02TP Study_Infants_Selected dose (Experimental): Infants who received 2 doses of the altSonflex1-2-3 vaccine on Day 1 and Day 169 in the H06_02TP parent study.
  Interventions: Biological: AltSonflex1-2-3
- H06_02TP Study_ Infants_Control (Active Comparator): Infants who received 1 dose of the TYPHIBEV vaccine on Day 1 and 1 dose of the Infanrix hexa vaccine on Day 169 in the H06_02TP parent study.
  Interventions: Biological: Infanrix hexa; Biological: TYPHIBEV

INTERVENTIONS:
Biological: AltSonflex1-2-3 — No intervention is administered in this extension study. The selected dose of altSonflex1-2-3 vaccine was administered intramuscularly in the participants' thigh during the H06_01TP (212149) parent study on Day 1, Day 85, and Day 253; or on Day 1 and Day 169 during the H06_02TP (219449) study.
  Other Names: GSK's Shigella vaccine
  Arms: H06_01TP Study_Infants_Selected dose; H06_02TP Study_Infants_Selected dose
Biological: Menveo — No intervention is administered in this extension study. The Menveo vaccine was administered intramuscularly in the participants' thigh on Day 1 and Day 85 during the H06_01TP (212149) parent study.
  Other Names: GSKs Meningococcal A, C, Y and W-135 conjugate vaccine
  Arms: H06_01TP Study_ ST2_Infants_Control
Biological: Infanrix hexa — No intervention is administered in this extension study. The Infanrix hexa vaccine was administered intramuscularly in the participants' thigh on Day 281 during the H06_01TP (212149) study; or on Day 169 during the H06_02TP (219449) parent study.
  Other Names: GSKs Diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis (inactivated), and Haemophilus influenzae type b vaccine
  Arms: H06_01TP Study_ ST2_Infants_Control; H06_02TP Study_ Infants_Control
Biological: TYPHIBEV — No intervention is administered in this extension study. The TYPHIBEV vaccine was administered intramuscularly in the participants' thigh on Day 1 during the H06_02TP (219449) parent study.
  Other Names: Biological E. Limiteds Typhoid Vi-CRM197 conjugate vaccine
  Arms: H06_02TP Study_ Infants_Control

SUMMARY:
The current study is a follow-up to 2 previous parent studies, a dose-selection study with 3 different dose-levels of the altSonflex1-2-3 vaccine in a schedule of 3 vaccinations (H06_01TP study [NCT05073003, 212149]) and a study with an alternate 2 vaccination schedule H06_02TP study [NCT06663436, 219449]). The current study aims to assess the longevity of the immune response to the selected dose of the altSonflex1-2-3 vaccine 1, 2, and 3 years after the last vaccination in African children. The study involves no new vaccinations but will collect immunogenicity blood samples from participants.

ELIGIBILITY:
Inclusion Criteria:

* Children who, as infants, previously participated in two completed studies (H06_01TP or H06_02TP) and were vaccinated with 3 or 2 doses of altSonflex1-2-3 or control vaccines, respectively, completed all previous vaccinations and are 12±1 months after the last altSonflex1-2-3 vaccination.
* Individuals in good health as determined by medical history since last study visit and clinical judgment of the investigator.

Exclusion Criteria:

* Serious and significant progressive, unstable, or uncontrolled clinical condition(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* Clinical condition(s) representing a contraindication to blood draws.
* Any behavioural or cognitive impairment or psychiatric disease.
* Acute disease and/or fever at the time of enrollment.
* Individuals with known or suspected HIV infection or HIV-related disease, with history of an autoimmune disorder or any other known or suspected impairment/alteration of the immune system, or under immunosuppressive therapy.
* Receipt of immunoglobulins and/or any blood products or plasma derivatives, during the period starting 3 months before each study visit.

Ages: 26 Months to 55 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 528 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Anti-serotype specific Shigella lipopolysaccharide (LPS)/O-antigen (OAg) serum immunoglobulin G (IgG), as measured by GVGH enzyme-linked immunosorbent assay . (ELISA) | At Visit 1 of the current study (12 months after last vaccination in the parent studies)
  S. sonnei, S. flexneri 1b, S. flexneri 2a, and S. flexneri 3a serotypes will be tested.
Anti-serotype specific Shigella LPS/OAg serum IgG, as measured by GVGH ELISA | At Visit 2 of the current study (24 months after last vaccination in the parent studies)
  S. sonnei, S. flexneri 1b, S. flexneri 2a, and S. flexneri 3a serotypes will be tested.
Anti-serotype specific Shigella LPS/OAg serum IgG, as measured by GVGH ELISA | At Visit 3 of the current study (36 months after last vaccination in the parent studies)
  S. sonnei, S. flexneri 1b, S. flexneri 2a, and S. flexneri 3a serotypes will be tested.

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf